CLINICAL TRIAL: NCT06748781
Title: Clinical and Radiographic Evaluation of Calcium Hypochlorite Versus Saline As Root Canal Irrigants in Pulpectomy of Primary Molars: a Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmine Abdo Helmy ElAssar, Yasmine Abdo Helmy ElAssar, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ca(OCl)2 Irrigation
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Irreversible Pulpitis
Keywords: calcium hypochlorite; irrigation; saline; irreversible pulpitis; calcium hydroxide with iodoform; primary molars; post operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Root Canal Irrigants

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- • Pulpectomy using Calcium Hypochlorite 2.5% as root canal irrigant (Experimental): Pulpectomy using 2.5% Calcium Hypochlorite root canal irrigant
  Interventions: Procedure: Pulpectomy using 2.5% Calcium Hypochlorite root canal irrigant.
- • Pulpectomy using Saline as root canal irrigant (Active Comparator): Pulpectomy using Saline as root canal irrigant.
  Interventions: Procedure: Pulpectomy using Saline as root canal irrigant

INTERVENTIONS:
Procedure: Pulpectomy using 2.5% Calcium Hypochlorite root canal irrigant. — 2.5% Calcium Hypochlorite used as root canal irrigant during the pulpectomy procedure in mandibular primary molars.
  Other Names: 2.5% Ca(OCl)2 Pulpectomy
  Arms: • Pulpectomy using Calcium Hypochlorite 2.5% as root canal irrigant
Procedure: Pulpectomy using Saline as root canal irrigant — Saline used as root canal irrigant during the pulpectomy procedure in mandibular primary molars.
  Other Names: Saline Pulpectomy
  Arms: • Pulpectomy using Saline as root canal irrigant

SUMMARY:
The aim of this study is to evaluate the clinical and radiographic success of Calcium Hypochlorite versus Saline as root canal irrigants in pulpectomy of primary molars.

The research question it aims to answer is:

In pulpectomy of primary molars will the use of calcium hypochlorite as root canal irrigant result in superior clinical and radiographic success to saline?

DETAILED DESCRIPTION:
Dental caries is a progressive disease of the dental hard tissue that may lead to pulpal, periapical, and/or intraradicular infections if not managed in its initial stages. Treating caries in primary dentition is necessary to prevent the spread of bacteria, infection of the pulp, abscess, or facial cellulitis and to maintain tooth space.

The operator can choose the most appropriate treatment, including pulpotomy, pulpectomy, direct pulp capping, or indirect pulp capping, according to the child's signs and symptoms, pulp vitality, and radiographic evaluation.

Pulpectomy procedure involves the removal of the entire pulp tissue from the crown and root canals. Proper instrumentation, irrigation, and root canal obturation are all necessary for a successful pulpectomy. Root canal irrigants are essential for cleaning the root canal system, dissolving tissues, and removing the debris. Therefore, the choice of suitable root canal irrigant is important for the success of pulpectomy treatment.

Saline has been commonly used as a root canal irrigant for pulpectomy of primary molars with irreversible pulpitis; however, it only provides lubrication and cleaning actions without any tissue dissolving or disinfecting properties.

(Nelson-Filho et al., 2018) conducted a study to compare the bacterial contamination identified in the root canals of primary teeth with irreversible inflammatory pulpitis and in teeth showing apical periodontitis. The findings showed that there is almost always bacterial contamination of pulp tissue of primary teeth with irreversible pulpitis whenever the cause is carious pulp exposure.

In a study conducted by (Walia et al., 2019) four irrigation solutions (2% chlorhexidine, 1% NaOCl, saline, and laser irradiation) were compared. It was found that all three irrigation solutions, with the exception of saline, were successful in lowering the microbial count.

Compared to saline, Ca(OCl)2 has significant tissue dissolving and high antibacterial properties sufficient to ensure successful root canal pulpectomy.

It was demonstrated that the cytotoxicity of Ca(OCl) is time and dose-dependent manner. Another study by Blattes et al., 2017 illustrated that Ca(OCl)2 showed favorable results of cell viability and a low-level inflammatory response. Ca(OCl)2 showed acceptable cytotoxicity and biocompatibility as a root canal irrigant.

Rationale Calcium Hypochlorite (Ca(ClO)2) is used for water purification and has been suggested to be used in endodontics due to its capacity for tissue dissolution and its antimicrobial properties which is almost comparable to that of NaOCl and exhibit less cytotoxicity than NaOCl.

Up to our knowledge, no clinical trials in the literature have been done to compare the clinical and radiographic success of Calcium Hypochlorite versus Saline as root canal irrigant in pulpectomy of primary molars. Thus, the purpose of the present study is to investigate the clinical and radiographic success of these two materials.

* The benefits of this study to the participants:

  1. Better anti-microbial efficacy.
  2. Good tissue tolerance.
* The benefits of this study to the population:

Improving the quality of life for the patients by providing successful treatment with less post-operative complications.

•The benefits of this study to the clinicians:

1. Providing a novel and alternative treatment option.
2. Less post-operative complications.
3. Simplicity in the preparation and less cost by obtaining a universal root canal irrigant that can manage all cases of primary teeth that need pulp therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Criteria:

   * Children aged between 4 years and 7 years.
   * Mandibular primary molars with deep caries lesion involving pulp.
   * Mandibular primary molars that exhibit symptoms of irreversible pulpitis.
   * Normal gingival and periodontal condition, with no sensitivity to vestibular palpation, and no pain on percussion test.
   * No history of swelling, fistula or sinus tract related to the offending molar.
2. Radiographic criteria:

   * No sign of radiolucency in periapical or furcation area.
   * No widening of PDL space or loss of lamina dura continuity.
   * No evidence of internal/external pathologic root resorption.

Exclusion Criteria:

* Uncooperative children to avoid time waste and attrition bias.
* Children with systemic disease as some systemic diseases may have effect on the outcome (Segura-Egea et al., 2023).
* Lack of informed consent by the child patient's parent to be approved ethically.
* Unable to attend follow-up visits to avoid attrition bias by decreasing number of drop off cases.
* Refusal of participation as the parent of child has the authority of participation.
* Teeth near exfoliation time showing root resorption.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Absence of post-operative pain. | 1-week changes from baseline pulp condition
  Asking the patient and/or guardian. Outcome measuring unit: Binary (Yes/No)

SECONDARY OUTCOMES:
Absence of Swelling/Sinus or Fistula. | at 3,6,9 and 12 months changes from the baseline pulp condition.
  Visual clinical examination. Outcome measuring unit: Binary (yes/no)
Absence of Pain to percussion | at 3,6,9 and 12 months changes from the baseline pulp condition.
  Percussion test using the back of a dental mirror. Outcome measuring unit :Binary (yes/no)
Pathologic mobility | at 3,6,9 and 12 months changes from the baseline pulp condition.
  Mobility test (pressure using the end of two dental mirrors). Outcome measuring unit :Binary (yes/no)
Absence of furcation or periapical radiolucency. | at 6 and 12 months changes from the baseline pulp condition.
  Intraoral digital periapical X-ray. Outcome measuring unit :Binary (present/absent)
Absence of external or internal root resorption. | at 6 and 12 months changes from the baseline pulp condition.
  Intraoral digital periapical X-ray. Outcome measuring unit :Binary (yes/no)
Widening of periodontal membrane space | at 6 and 12 months changes from the baseline pulp condition.
  Intraoral digital periapical X-ray. Outcome measuring unit :Binary (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Educational Dental Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided